CLINICAL TRIAL: NCT04808622
Title: Randomized, Double-blind, Placebo-controlled, Pharmacokinetic, Pharmacodynamic Study of Trans Sodium Crocetinate Utilizing Transcutaneous Oximetry Measurement in Healthy Volunteers
Brief Title: Safety and Efficacy of Trans Sodium Crocetinate (TSC) in Enhancing Tissue Oxygen Levels in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 200-301
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-08

CONDITIONS: Healthy Subjects
Keywords: Transcutaneous oximetry
MeSH Terms: interventions — trans-sodium crocetinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TSC 0.5 mg/kg (Experimental): TSC 0.5 mg/kg given as a one-time IV bolus injection
  Interventions: Drug: Trans-Sodium Crocetinate
- TSC 1.0 mg/kg (Experimental): TSC 1.0 mg/kg given as a one-time IV bolus injection
  Interventions: Drug: Trans-Sodium Crocetinate
- TSC 1.5 mg/kg (Experimental): TSC 1.5 mg/kg given as a one-time IV bolus injection
  Interventions: Drug: Trans-Sodium Crocetinate
- TSC 2.0 mg/kg (Experimental): TSC 2.0 mg/kg given as a one-time IV bolus injection
  Interventions: Drug: Trans-Sodium Crocetinate
- TSC 2.5 mg/kg (Experimental): TSC 2.5 mg/kg given as a one-time IV bolus injection
  Interventions: Drug: Trans-Sodium Crocetinate
- Placebo (Placebo Comparator): 7 mL normal saline given as a one-time IV bolus injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trans-Sodium Crocetinate — TSC given as a one-time IV bolus injection
  Other Names: TSC
  Arms: TSC 0.5 mg/kg; TSC 1.0 mg/kg; TSC 1.5 mg/kg; TSC 2.0 mg/kg; TSC 2.5 mg/kg
Drug: Placebo — Placebo normal saline given as a one-time 7 mL one-time IV bolus injection
  Other Names: 0.9% Sodium Chloride (NaCl)
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, pharmacokinetic, pharmacodynamic study.

Subjects will be randomized to TSC or placebo to determine the effect of Trans Sodium Crocetinate (TSC) on Transcutaneous Oximetry Measurements (tcpO2) following a single administration of TSC in subjects breathing oxygen (O2).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, pharmacokinetic, pharmacodynamic study of Trans Sodium Crocetinate (TSC) in healthy volunteers. The primary objective is to determine the effect of TSC on transcutaneous oximetry measurements (tcpO2) following a single administration of TSC in subjects breathing oxygen (O2).

30 healthy volunteers will be randomized to one of 6 treatment groups, to include 5 TSC doses (0.5, 1.0, 1.5, 2.0, and 2.5 mg/kg) and placebo normal saline (7 mL). TcpO2 sensors will be applied to 4 standardized areas on the lower extremity. Subjects will be placed on O2 via simple face mask at 6 L/minute, and will remain on O2 for 70 minutes prior to study drug administration. The first 10 minutes will allow for equilibration of O2 levels, and the subsequent 60 minutes will serve as the baseline period. TcpO2 values and SpO2 will be recorded every 5 minutes during the above periods. At the end of the 70-minute equilibration/baseline period, subjects will receive a single IV bolus injection of TSC at a dose of 0.5, 1.0, 1.5, 2.0 or 2.5 mg/kg, or placebo. Study drug will be administered in a blinded fashion.

After study drug is administered, subjects will continue on O2 and be evaluated for an additional 60 minutes, with tcpO2 and SpO2 recorded at 1, 2, and 5 minutes post-dose, and every 5 minutes thereafter.

Prior to and following study drug administration, PK samples will be obtained pre-dose, and 1, 10, 30, and 90 minutes post-dose.

After the 60 minute post-treatment evaluation period, oxygen will be discontinued and the tcpO2 sensor electrodes removed. Subjects will remain in the procedure room for an additional 30 minutes to allow for collection of the 1.5-hour PK blood draw and repeat vital signs. Subjects will remain in the clinic overnight for observation and discharged the following morning.

Subjects will be contacted by telephone at 48 hours (+ 2 days) for a safety follow up to assess adverse events and new medications.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18-50
2. Able and willing to lie quietly supine or semi-recumbent for up to 2.5 hours
3. Abstinence from exercise, caffeine, alcohol, nicotine, and a heavy meal prior to testing on the day of the Treatment Visit
4. Subject is able to communicate effectively with the Investigator and to comply with all study requirements, restrictions, and directions from the study staff
5. Females of childbearing potential must have a negative blood pregnancy test at screening and agree to use one of the accepted contraceptive regimens, or a double method of birth control (e.g. condom and spermicide), during the study and at least 30 days after the last dose of study drug. Females of non-childbearing potential should be surgically sterile or at least one year post-menopausal.
6. Males who engage in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g. condom and spermicide) and agree not to donate sperm during the study and for at least 90 days after the last dose of study drug

Exclusion Criteria:

1. Allergy to study medication
2. Pregnant or breastfeeding
3. Current smoker and/or any nicotine use within 4 hours of the start of tcpO2 procedures, to include e-cigarette vaping, snuff, chew, nicotine gum and nicotine patches
4. Body Mass Index (BMI) > 30
5. Positive test results for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg), or Hepatitis C Antibody (HCVAb)
6. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening
7. Plasma donation within 7 days prior to screening
8. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening
9. Any skin condition on limbs to be tested that could impair testing (rash, wound, prior radiation therapy, other skin conditions, per Principal Investigator (PI) discretion)
10. Known cardiovascular disease, including treated or untreated hypertension
11. Significant respiratory disease and/or any other significant medical condition
12. Subject has an acute illness (gastrointestinal infection, influenza, or known inflammatory process) at the Treatment Visit
13. Urine screen positive for drugs or positive breathalyzer for alcohol (at screening and enrollment)
14. Concomitant medications used to treat a diagnosed medical condition
15. Subject who, for any reason, is deemed by the Investigator to be unsuitable for the study; or has any condition that would interfere with the evaluation of tissue oxygen measurements or PK of the investigational drug; or is otherwise unable to comply with the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Kankam, MD, PhD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas Inc, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TSC 0.5 mg/kg | TSC 1.0 mg/kg | TSC 1.5 mg/kg | TSC 2.0 mg/kg | TSC 2.5 mg/kg | Placebo
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TSC 0.5 mg/kg | TSC 1.0 mg/kg | TSC 1.5 mg/kg | TSC 2.0 mg/kg | TSC 2.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 5 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (10.93) | 37.4 (11.44) | 33.0 (9.17) | 29.8 (5.12) | 40.4 (8.41) | 27.0 (5.00) | 33.1 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 2 | 3 | 1 | 14
  Male | 3 | 2 | 2 | 3 | 2 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 3 | 5 | 4 | 4 | 5 | 5 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 3 | 3 | 3 | 4 | 19
  White | 2 | 1 | 2 | 1 | 2 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Summary of ANOVA Results (Difference [95% Confidence Interval]) for tcpO2 Time-Matched Values by TSC Cohort Compared to Placebo.
Description: Determine the Dose-Response of TSC on tcpO2 Following a Single Administration of TSC in Subjects Breathing O2.
Time Frame: 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 minutes post-dose
Population: This analysis is a comparison of TSC cohort compared to Placebo; therefore, the total number analyzed is less, as there are not specific data reported for the Placebo cohort. One subject from the TSC 2.5 mg/kg cohort was excluded due to subcutaneous injection of TSC.
Measure: Number (95% Confidence Interval); unit: mmHg
Arm/Group | TSC 0.5 mg/kg | TSC 1.0 mg/kg | TSC 1.5 mg/kg | TSC 2.0 mg/kg | TSC 2.5 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4
mmHg
  0-5 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  0-5 Minutes Post-Dose | -4.1 [-37.0 to 28.7] | -7.6 [-41.1 to 25.9] | -3.3 [-36.1 to 29.5] | 10.5 [-22.4 to 43.3] | 21.1 [-13.7 to 55.9]
  5-10 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  5-10 Minutes Post-Dose | 5.6 [-27.2 to 38.4] | 2.7 [-30.8 to 36.2] | 0.5 [-32.3 to 33.4] | 19.2 [-13.6 to 52.0] | 37.0 [2.2 to 71.9]
  10-15 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  10-15 Minutes Post-Dose | 20.2 [-12.6 to 53.0] | 8.2 [-25.3 to 41.7] | 11.4 [-21.5 to 44.2] | 11.2 [-21.7 to 44.0] | 37.2 [2.3 to 72.0]
  15-20 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  15-20 Minutes Post-Dose | 18.6 [-14.3 to 51.4] | 19.0 [-14.5 to 52.5] | 13.4 [-19.4 to 46.2] | 16.4 [-16.4 to 49.2] | 29.8 [-5.1 to 64.6]
  20-25 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  20-25 Minutes Post-Dose | 11.1 [-21.7 to 44.0] | 22.9 [-10.6 to 56.4] | 14.8 [-18.0 to 47.6] | 16.2 [-16.7 to 49.0] | 34.9 [0.0 to 69.7]
  25-30 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  25-30 Minutes Post-Dose | 13.6 [-19.3 to 46.4] | 24.3 [-9.2 to 57.8] | 10.2 [-22.6 to 43.0] | 7.1 [-25.7 to 40.0] | 26.1 [-8.8 to 60.9]
  30-35 Minutes Post-Dose: number analyzed (Participants) | 5 | 4 | 5 | 5 | 4
  30-35 Minutes Post-Dose | 9.6 [-23.3 to 42.4] | 13.6 [-19.9 to 47.1] | 8.2 [-24.7 to 41.0] | 0.1 [-32.8 to 32.9] | 20.9 [-13.9 to 55.7]
  35-40 Minutes Post-Dose | 11.6 [-21.3 to 44.4] | 33.3 [0.5 to 66.1] | 14.4 [-18.4 to 47.2] | 3.1 [-29.7 to 35.9] | 26.0 [-8.8 to 60.9]
  40-45 Minutes Post-Dose | 14.7 [-18.1 to 47.5] | 43.5 [10.7 to 76.3] | 14.9 [-17.9 to 47.7] | 6.9 [-25.9 to 39.7] | 23.6 [-11.3 to 58.4]
  45-50 Minutes Post-Dose | 15.8 [-17.1 to 48.6] | 26.4 [-6.4 to 59.2] | 17.4 [-15.4 to 50.2] | 4.8 [-28.0 to 37.7] | 24.1 [-10.8 to 58.9]
  50-55 Minutes Post-Dose | 3.7 [-29.1 to 36.5] | 4.4 [-28.4 to 37.2] | 6.2 [-26.6 to 39.0] | -3.3 [-36.2 to 29.5] | 16.1 [-18.7 to 50.9]
  55-60 Minutes Post-Dose | 12.4 [-20.4 to 45.3] | 18.1 [-14.7 to 51.0] | 9.0 [-23.8 to 41.8] | 12.7 [-20.1 to 45.5] | 28.7 [-6.1 to 63.5]

2. Primary Outcome: Determine the Dose-Response of TSC on tcpO2 Following a Single Administration of TSC in Subjects Breathing O2.
Description: Summary Statistics of tcpO2 Levels (mmHg) Overall Measurements (Median of 4 Sensors) in Healthy Subjects
Time Frame: 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 minutes post-dose
Population: One subject from the TSC 2.5 mg/kg cohort was excluded due to subcutaneous injection of TSC.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Placebo given as a one-time IV bolus injection
Arm/Group | TSC 0.5 mg/kg | TSC 1.0 mg/kg | TSC 1.5 mg/kg | TSC 2.0 mg/kg | TSC 2.5 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 5
mmHg
  Baseline 0 to 5 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 0 to 5 Minutes (Period 1) | 175.3 (65.82) | 153.1 (41.18) | 178.0 (62.28) | 179.9 (44.78) | 162.4 (60.01) | 197.2 (35.64)
  0 to 5 Minutes (Period 2) | 165.1 (74.19) | 165.8 (41.36) | 180.0 (46.72) | 203.3 (51.59) | 194.7 (104.76) | 212.2 (42.48)
  0 to 5 Minutes (Period 2-Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  0 to 5 Minutes (Period 2-Period 1) | 11.2 (18.56) | 5.6 (10.79) | 12.1 (16.57) | 25.8 (20.66) | 36.4 (45.84) | 15.4 (10.74)
  Baseline 5 to 10 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 5 to 10 Minutes (Period 1) | 185.2 (72.12) | 159.4 (40.33) | 179.8 (60.77) | 187.4 (46.58) | 160.1 (53.88) | 201.3 (34.41)
  5 to 10 Minutes (Period 2) | 170.0 (77.42) | 159.4 (41.05) | 184.1 (57.54) | 206.9 (52.15) | 194.0 (112.18) | 191.4 (29.89)
  5 to 10 Minutes (Period 2 - Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  5 to 10 Minutes (Period 2 - Period 1) | 9.5 (15.92) | 4.3 (5.10) | 4.4 (4.88) | 23.1 (22.02) | 40.9 (57.17) | 3.9 (8.61)
  Baseline 10 to 15 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 10 to 15 Minutes (Period 1) | 180.0 (80.42) | 160.3 (36.89) | 176.2 (56.77) | 196.6 (48.62) | 162.6 (52.24) | 209.1 (38.36)
  10 to 15 Minutes (Period 2) | 170.6 (81.23) | 167.5 (47.82) | 183.9 (48.67) | 201.8 (22.56) | 197.6 (113.49) | 189.5 (33.80)
  10 to 15 Minutes (Period 2 - Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  10 to 15 Minutes (Period 2 - Period 1) | 22.2 (38.11) | 7.9 (12.62) | 13.3 (12.05) | 13.1 (18.02) | 39.1 (62.75) | 2.0 (4.36)
  Baseline 15 to 20 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 15 to 20 Minutes (Period 1) | 178.6 (73.05) | 162.3 (36.34) | 180.7 (64.26) | 200.9 (51.63) | 172.8 (65.31) | 211.9 (38.92)
  15 to 20 Minutes (Period 2) | 172.9 (81.80) | 174.8 (51.85) | 184.5 (43.30) | 206.4 (20.96) | 197.8 (110.08) | 191.3 (35.59)
  15 to 20 Minutes (Period 2 - Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  15 to 20 Minutes (Period 2 - Period 1) | 18.6 (34.55) | 16.8 (22.89) | 13.4 (14.46) | 16.4 (17.44) | 29.8 (45.52) | 0.0 (0.00)
  Baseline 20 to 25 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 20 to 25 Minutes (Period 1) | 190.9 (74.50) | 164.8 (29.95) | 173.2 (55.79) | 202.8 (46.65) | 173.4 (64.31) | 216.6 (37.24)
  20 to 25 Minutes (Period 2) | 171.0 (82.54) | 180.6 (57.06) | 180.2 (46.04) | 214.4 (41.19) | 204.1 (113.93) | 196.3 (47.51)
  20 to 25 Minutes (Period 2 - Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  20 to 25 Minutes (Period 2 - Period 1) | 11.2 (18.64) | 20.7 (38.43) | 14.8 (14.47) | 16.2 (15.83) | 34.9 (49.62) | 0.0 (0.00)
  Baseline 25 to 30 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 25 to 30 Minutes (Period 1) | 190.5 (78.11) | 166.4 (31.95) | 178.8 (59.96) | 200.8 (44.50) | 180.1 (73.41) | 216.2 (34.75)
  25 to 30 Minutes (Period 2) | 171.9 (84.09) | 182.0 (64.23) | 182.0 (44.54) | 202.7 (36.80) | 202.0 (116.66) | 184.8 (48.54)
  25 to 30 Minutes (Period 2 - Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  25 to 30 Minutes (Period 2 - Period 1) | 13.6 (25.57) | 22.1 (44.13) | 10.2 (14.06) | 7.2 (7.91) | 26.1 (42.86) | 0.0 (0.00)
  Baseline 30 to 35 Minutes (Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  Baseline 30 to 35 Minutes (Period 1) | 184.5 (76.58) | 148.1 (38.63) | 175.8 (64.14) | 212.1 (46.47) | 175.4 (74.39) | 207.9 (27.97)
  30 to 35 Minutes (Period 2) | 167.0 (87.89) | 172.4 (51.69) | 176.8 (41.05) | 200.5 (37.18) | 198.0 (117.16) | 186.9 (51.28)
  30 to 35 Minutes (Period 2 - Period 1): number analyzed (Participants) | 5 | 4 | 5 | 5 | 4 | 5
  30 to 35 Minutes (Period 2 - Period 1) | 15.4 (32.38) | 17.3 (26.50) | 14.0 (20.96) | 5.9 (11.59) | 26.8 (42.32) | 5.9 (13.08)
  Baseline 35 to 40 Minutes (Period 1) | 182.4 (68.80) | 151.5 (37.51) | 175.5 (61.35) | 217.9 (55.35) | 177.8 (73.80) | 217.0 (38.14)
  35 to 40 Minutes (Period 2) | 170.3 (93.45) | 180.9 (66.13) | 177.4 (38.83) | 200.3 (40.66) | 200.8 (122.86) | 180.7 (56.25)
  35 to 40 Minutes (Period 2 - Period 1) | 12.7 (21.04) | 34.5 (47.14) | 15.6 (15.71) | 4.3 (9.50) | 27.2 (49.34) | 1.2 (2.57)
  Baseline 40 to 45 Minutes (Period 1) | 188.5 (63.41) | 141.3 (35.52) | 178.6 (58.66) | 208.2 (61.65) | 181.6 (81.21) | 210.5 (38.04)
  40 to 45 Minutes (Period 2) | 176.2 (92.17) | 180.6 (66.93) | 174.3 (35.85) | 209.2 (52.68) | 199.8 (127.19) | 179.0 (58.21)
  40 to 45 Minutes (Period 2 - Period 1) | 14.7 (26.44) | 43.5 (70.00) | 14.9 (16.14) | 6.9 (9.61) | 23.6 (45.97) | 0.0 (0.00)
  Baseline 45 to 50 Minutes (Period 1) | 181.8 (71.14) | 148.9 (34.66) | 177.1 (61.65) | 208.7 (59.68) | 182.5 (87.39) | 210.0 (38.80)
  45 to 50 Minutes (Period 2) | 178.5 (94.21) | 173.4 (58.98) | 170.1 (39.37) | 211.1 (53.79) | 204.6 (119.52) | 177.3 (63.38)
  45 to 50 Minutes (Period 2 - Period 1) | 16.6 (28.69) | 27.2 (56.55) | 18.2 (17.92) | 5.7 (12.36) | 24.9 (31.39) | 0.8 (1.79)
  Baseline 50 to 55 Minutes (Period 1) | 180.7 (72.77) | 168.9 (49.20) | 181.7 (56.10) | 211.6 (49.69) | 183.3 (97.50) | 200.5 (32.29)
  50 to 55 Minutes (Period 2) | 173.2 (91.33) | 174.4 (60.55) | 178.2 (40.18) | 208.1 (50.63) | 203.6 (114.20) | 181.2 (68.49)
  50 to 55 Minutes (Period 2 - Period 1) | 10.3 (16.19) | 11.0 (14.14) | 12.8 (12.81) | 3.3 (4.10) | 22.7 (18.62) | 6.6 (14.76)
  Baseline 55 to 60 Minutes (Period 1) | 171.9 (70.80) | 160.8 (45.32) | 177.2 (47.41) | 196.9 (43.77) | 179.0 (84.54) | 202.1 (35.29)
  55 to 60 Minutes (Period 2) | 172.5 (93.64) | 175.5 (69.98) | 172.1 (42.22) | 209.9 (50.43) | 205.9 (119.43) | 174.7 (65.35)
  55 to 60 Minutes (Period 2 - Period 1) | 13.5 (24.05) | 19.2 (32.20) | 10.1 (14.00) | 13.8 (10.39) | 29.8 (31.53) | 1.1 (2.35)

ADVERSE EVENTS:
Time Frame: AEs were collected up to 5 days from the start of equilibration (Day 0) through the 48-hour follow-up visit (Day 3 +2d).
Arm/Group | TSC 0.5 mg/kg | TSC 1.0 mg/kg | TSC 1.5 mg/kg | TSC 2.0 mg/kg | TSC 2.5 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 2/5 | 3/5 | 1/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSC 0.5 mg/kg (N=5) | TSC 1.0 mg/kg (N=5) | TSC 1.5 mg/kg (N=5) | TSC 2.0 mg/kg (N=5) | TSC 2.5 mg/kg (N=5) | Placebo (N=5)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Streaking (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post-Procedural Erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post-Procedural Pruritus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of this study include the small sample size and the observed variability across individual TcpO2 sensors that did not allow for pooling of sensor readings for a direct time-matched comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT04808622/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT04808622/SAP_001.pdf